CLINICAL TRIAL: NCT02225782
Title: A Randomized Double-blind Controlled Study to Compare the Effectiveness of 1.0 Versus 2.0 mg Alteplase (tPA) Dosing in Restoring
Brief Title: Trial to Compare 1.0 Versus 2.0 mg Alteplase (tPA) Dosing in Restoring Hemodialysis Catheter Function
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Windsor (Other)
Collaborators: The Kidney Foundation of Canada (Other)
Responsible Party: Principal Investigator, Maher M. El-Masri, Professor and Faculty Research Chair, University of Windsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KFOC140002
Record Dates: First submitted 2014-08-22; First posted 2014-08-26 (Estimated); Last update posted 2016-05-12 (Estimated); Status verified 2016-05

CONDITIONS: Kidney Disease
Keywords: Alteplase; Hemodialysis Catheter; Occlusion; Renal Failure
MeSH Terms: conditions — Kidney Diseases; Bites and Stings; Renal Insufficiency | interventions — Tissue Plasminogen Activator

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1.0 mg alteplase (tPA) (Active Comparator): 1.0 mg tPA to be injected at the catheter site for a maximum of 3 repeats if the catheter site occlusion is not resolved with 30 minute wait between each repeat
  Interventions: Drug: Alteplase
- 2.0 mg alteplase (tPA) (Experimental): 2.0 mg tPA to be injected at the catheter site for a maximum of 3 repeats if the catheter site occlusion is not resolved with 30 minute wait between each repeat
  Interventions: Drug: Alteplase

INTERVENTIONS:
Drug: Alteplase — Alteplase is a fibrinolytic drug widely used to restore hemodialysis catheter patency.
  Other Names: tPA

SUMMARY:
Hemodialysis is a procedure that kidney physicians perform when the kidneys fail and can no longer clean the blood and remove extra fluid and toxins from the body. Hemodialysis therefore requires access to reach the blood through either a surgically created permanent fistula or graft or through the insertion of a temporary catheter in one of the large body veins. While the use of fistulas or grafts is preferred because they are permanent, there may be conditions that prevent patients from having them and a hemodialysis catheter may be used instead. The problem with the use of catheters however is that they can become blocked due to the formation of blood clots. Kidney physicians try to resolve occlusion of hemodialysis catheters by injecting a medication called Alteplase which breaks the clot at the catheter site. There is no consensus in the medical community as to how much of the medication should be injected at the occluded catheter site. While some kidney physicians and studies recommend the use of 1.0 mg of the medication at each occlusion site, others recommend that 2.0 mg of the medication should be used. Thus, the purpose of this randomized clinical trial is to compare the effectiveness of 1.0mg versus 2.0mg dose of alteplase in resolving blood clots in hemodialysis catheters.

The investigators will recruit patients for the study from a regional hemodialysis unit that is located in southwestern Ontario. Patients who agree to participate in this research and experiences occlusion of their hemodialysis catheters will be divided into two groups; making sure that this division is completely by chance. The first group will receive 1.0mg alteplase, while the second will receive 2.0mg Alteplase. The investigators will collect information on both groups and will run statistical analysis of these information to compare the results of clot resolution between the groups.

DETAILED DESCRIPTION:
Objectives The primary purpose of this study is to examine the effectiveness of tPA 2.0 mg as compared to 1.0 mg in restoring hemodialysis catheter (HDC) function after blood occlusion.

Specifically, the study aims to:

1. Examine the risk reduction (absolute and relative) in HDC occlusion that is associated with the administration of 2.0mg tPA as opposed to 1.0 mg tPA in HD patients
2. Compare the median catheter removal time between hemodialysis (HD) patients who experienced HDC occlusion and were managed with tPA 2.0 mg and those who were managed with tPA 1.0 mg.
3. Compare the average number of tPA repeats between HD patients who receive 2.0 mg and those who receive 1.0 mg dose.
4. Compare the rate of HDC stripping between HD patients who experienced HDC occlusion and were managed with 2.0 mg tPA and those who were managed with 1.0 mg tPA.

Hypotheses

1. Patients who receive tPA 2.0 mg dose for the management of their HDC blood occlusion will experience a higher rate of HDC function restoration than patients who receive tPA 1.0 mg dose.
2. Median time to HDC catheter removal after successful management of HDC occlusion with tPA will be higher among those who receive 2.0 mg tPA than those who receive 1.0 mg tPA.
3. b) The number of repeats of tPA administration will be less among patients who receive 2.0 mg dose than it is among those who receive 1.0 mg dose.
4. The rate of HDC stripping for HD patients who experienced catheter occlusion will be lower among patients who received 2.0 mg tPA than it is among patients who received 1.0 mg tPA.

Methods and Materials

A double blind, randomized, controlled clinical trial will be conducted on consenting hemodialysis patients who will require tPA management of their HDC dysfunction. All patients will be recruited from a regional out-patient HD unit in southwestern Ontario. Eligible HD patients will be approached with verbal and written explanation about the research, and will be invited to sign a written consent to participate in the study. All consenting patients will be randomly assigned to either of the two study groups, based on allocation concealment principles, immediately after they experience HDC occlusion due to a blood clot. Patient recruitment will continue until a minimum sample of 75 participants per group is achieved, to provide a total minimum sample of 150 participants.

Recruitment Protocol All study participants will be recruited from the out-patient HD unit at our region, which provides HD services to an average of 250 patients at any given year. Prior to the initiation of the study, the research team will hold an information session to orient the staff at the HD unit to the study protocol. All HD patients who attend our regional unit will be approached with information about the study, its purpose and protocol, and will be asked to provide voluntary written consent to participate in the study. Consents will be sought from all prospective participants before an HDC occlusion takes place. Once an HDC occlusion is reported and the patient is deemed by the nurse to be eligible for tPA management according to the guidelines of the Medical Directive for tPA administration, the patient will be allocated to either of the study groups by a research assistant. Patient allocation will be performed based on a predetermined concealed random sequence to ensure that neither the patient nor members of the research team are aware of the patient random allocation to either of the study groups. To ensure that the two groups have an equal number of participants, block randomization approach with five participants per block will be implemented. In order to enhance the allocation concealment process, the random codes will be generated by a colleague who is not a member of the research team using a computer program. Each random allocation code will be kept according to the order of its sequence in an oblique envelope at a locked cabinet in the HD unit.

Data Collection and tPA Administration Protocols Once allocated to a treatment group, the patient will be blindly given the treatment according to the medical directive of the HD unit for the administration of tPA for the management of HDC occlusion. To ensure blinding of treatment, the two groups will be coded as "A" and "B" and these codes will only be known to the pharmacist (not involved with the study) who will pre-fill the tPA syringes and label them accordingly. Thus, the pharmacist will prepare all 1.0mg and the 2.0mg doses in 2.0ml syringes; whereby the 1.0mg dose will be prepared in a concentration of 1.0mg/2.0ml, while the 2.0mg dose will be prepared in a concentration of 2.0mg/2.0ml. The varying syringe concentrations will ensure that both doses are identical to ensure the blinding of the two study groups. Once ready to administer the tPA according to the medical directive, the HD nurse will instill the prefilled tPA solution into the occluded HDC lumen and allow it to dwell in the lumen for 30 minutes. The HD nurse will then withdraw 3.0 ml of blood from the occluded lumen and assess for patency. If there is a backflow and the HDC is deemed patent, the HD nurse will recommence HD. If the HDC lumen is not patent after the first instill, the HD nurse may repeat the tPA administration procedure up to a maximum of a total of three times before a referral for therapeutic radiology is arranged to strip the catheter. Data on the total number of repeats, the outcome of each repeat, and the outcome of the radiology will be collected. The nurse initiating the tPA medical directive will document the administration of tPA in the patient medication record according to their volume (i.e., 2ml pre-filled dose). He/she will also communicate the procedure to the Research Assistant for the study on a separate log book that will be kept at the nurses' station of the HD unit. The Research Assistant will review the log book on regular basis to collect data on the tPA administration procedure, demographic information, prognostic factors, participants' relevant medications and blood labs, and medical history. Patients will be followed up after tPA management until he/she reaches the study endpoint.

ELIGIBILITY:
Inclusion Criteria:

* A patient will be deemed eligible for inclusion in the study if he/she:

  1. Is ≥ 18 years of age,
  2. Is receiving HD for chronic renal failure using permanent HDC that is inserted in any of the following sites: internal jugular, subclavian, or femoral veins
  3. Has no medical contradiction for tPA management of partially or fully occluded HDC.

In addition, only the first occlusion event that requires tPA administration for a single catheter will be included. However, each new catheter insertion for the same patient during the study will be treated as a new event. That is, a single patient may be randomized more than one time if he/she experiences the insertion of more than one catheter during the course of the study

Exclusion Criteria:

* Pregnant women
* Patients who received ≤ 7 dialysis treatment sessions or have been on dialysis for less than 15 days
* Patients who had contraindications, allergies, or history of intolerances to tPA will be excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2014-10; Primary Completion 2016-07 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Restoration of hemodialysis catheter | 30 minutes after administration of the tPA at the catheter site
  The pharmacist will prepare all 1.0mg and the 2.0mg doses in 2.0ml syringes; whereby the 1.0mg dose will be prepared in a concentration of 1.0mg/2.0ml, while the 2.0mg dose will be prepared in a concentration of 2.0mg/2.0ml. The varying syringe concentrations will ensure that both doses are identical to ensure the blinding of the two study groups. Once ready to administer the tPA according to the medical directive, the HD nurse will instill the prefilled tPA solution into the occluded HDC lumen and allow it to dwell in the lumen for 30 minutes. The HD nurse will then withdraw 3.0 ml of blood from the occluded lumen and assess for patency. If there is a backflow and the HDC is deemed patent, the HD nurse will recommence HD. If the HDC lumen is not patent after the first instill, the HD nurse may repeat the tPA administration procedure up to a maximum of a total of three times before a referral for therapeutic radiology is arranged to strip the catheter

SECONDARY OUTCOMES:
Number of catheter strippings | after 3 repeates of tPA management with a waiting time of 30 minutes between each tPA repeat
  Comparing the number of catheter stripping procedures between patients who have their occluded catheters managed by 1.0 mg tPA versus 2.0 mg

CONTACTS AND LOCATIONS:
Overall Officials: Maher M El-Masri, PhD, Principal Investigator — University of Windsor; Albert Kadri, MD, Principal Investigator — Windsor Regional Hospital; Wasim S El Nekidy, PharmD, Principal Investigator — Windsor Regional Hospital
Locations (1):
- Windsor Regional Hospital, Windsor, Ontario, Canada